CLINICAL TRIAL: NCT04822116
Title: Continuation of Goal Directed Haemodynamic Optimization in the Postanaesthesia Care Unit on the Basis of Non-invasive Methods: a Randomized Controlled Trial.
Brief Title: Continuation of Goal Directed Haemodynamic Optimization in the PACU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, Clinical Professor, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IN-PACU-01
Record Dates: First submitted 2019-06-21; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Hemodynamic Instability; Postoperative Complications; Ultrasound Imaging
Keywords: Goal directed haemodynamic optimization; Ultrasound Imaging; Postoperative complications
MeSH Terms: conditions — Postoperative Complications | interventions — Crystalloid Solutions

STUDY DESIGN:
Intervention Model Description: In the study group volume therapy is based on variables like stroke volume and/or diameter of vena cava inferior based on a goal directed haemodynamic optimization protocol.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention): Standard of care defined as "standard operating procedure", including a goal directed intraoperative haemodynamic optimization protocol.
- goal directed intraoperative haemodynamic optimization (Active Comparator): Standard of care defined as "standard operating procedure", including a goal directed intraoperative haemodynamic optimization protocol. Additional application of a non-invasive haemodynamic optimization protocol in the post anaesthesia care unit.
  Interventions: Other: goal directed intraoperative haemodynamic optimization

INTERVENTIONS:
Other: goal directed intraoperative haemodynamic optimization — all interventions that were pre-specified to be administered as part of the protocol
  Other Names: crystalloids; transthoracic echocardiography; volume clamp method
  Arms: goal directed intraoperative haemodynamic optimization

SUMMARY:
Post-operative monitoring of all patients after anaesthesia in the post anaesthesia care unit (PACU) is standard of care today. It helps to reduce morbidity and even mortality in high-risk patients.

In addition to clinical monitoring by qualified staff, standard monitoring in the PACU includes non-invasive, intermittent, haemodynamic monitoring.

This research is going to investigate the influence of the continuation of goal directed haemodynamic optimization in the recovery room on the basis of non-invasive monitoring tools, i.e. ultrasound and the volume-clamp method, in regard of length of stay in the PACU and postoperative complications.

DETAILED DESCRIPTION:
Postoperative monitoring of all patients after surgery in post anaesthesia care unit (PACU) is standard of care today. It helps to reduce morbidity and even mortality in high-risk patients.

In addition to clinical monitoring by qualified staff, standard monitoring in the PACU includes non-invasive, intermittent, haemodynamic monitoring. The time of transfer of patients from the PACU to the general ward is assessed on the basis of several parameters. There is consensus on the most important endpoints of transferability: awareness, quality of spontaneous breathing, circulatory situation, bleeding situation, body temperature, diuresis and satisfactory freedom from pain and absence of nausea, but the processes and contents and how they can be established as quickly and sustainable as possible are not yet defined.

This research will investigate the influence of continuing non-invasive, goal-directed haemodynamic optimization in the recovery room, after major traumatological, general and vascular surgery.

In a randomized controlled trial the investigators will include a population of 80 patients with a minimum age of 18 years in the study after clarification and approval.

The control group will be routinely treated with an appropriate protocol for goal-oriented haemodynamic optimization. The study group will receive targeted haemodynamic optimization using Vigileo FlowTrac-Analysis and transthoracic echocardiography in the operation room and finger-cuff based pulse analysis technology in the PACU. The observed parameters of targeted haemodynamic optimization will be stroke volume and cardiac output, volume response parameters and collapsability of the inferior vena cava for the volume status.

As primary endpoints the investigators considered the number of postoperative complications. As secondary endpoints, the investigators will compare the time spent in the recovery room, the time spent in hospital and 28-day mortality and morbidity.

The hypothesis is that, in patients classified ASA II and III, a continuation of a targeted haemodynamic optimization in the PACU with non-invasive monitoring methods can reduce postoperative complications after a variety of surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA classification I-III undergoing abdominal surgery, surgery in urology or vascular surgery
* written consent

Exclusion Criteria:

* Age <18 years
* ASA classification IV or higher
* legal care relationship
* missing or faulty written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
acute kidney failure | through study completion, an average of 1 year
  Number of post-operative complications
pulmonary oedema | through study completion, an average of 1 year
  Number of post-operative complications
wound infection | through study completion, an average of 1 year
  Number of post-operative complications
pneumonia | through study completion, an average of 1 year
  Number of post-operative complications

SECONDARY OUTCOMES:
length of stay in the PACU | through study completion, an average of 1 year
  through study completion
length of stay in hospital | through study completion, an average of 1 year
  through study completion
28-day survival | through study completion, an average of 1 year
  through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, prof. Dr., Study Chair — University Hospital Schleswig-Holstein, Kiel
Locations (1):
- Universitätsklinikum Schleswig-Holstein Campus Kiel - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Deutschland (deu), Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldrete JA, Kroulik D A postanesthetic recovery score. Anesth Analg 1970; 49: 924-34. McLaren JM, Reynolds JA, Cox MM, et al. Decreasing the length of stay in phase I postanesthesia care unit: an evidence-based approach. J Perianesth Nurs 2015; 30: 116-23. Ameloot K, Van De Vijver K, Van Regenmortel N, et al. Validation study of Nexfin(R) continuous non-invasive blood pressure monitoring in critically ill adult patients. Minerva Anestesiol 2014; 80: 1294-301. Batz G, Dinkel M [Hemodynamic monitoring - imaging procedures / cardiac ultrasound]. Anasthesiol Intensivmed Notfallmed Schmerzther 2016; 51: 626-34. White PF, Song D New criteria for fast-tracking after outpatient anesthesia: a comparison with the modified Aldrete's scoring system. Anesth Analg 1999; 88: 1069-72. Broch O, Carstens A, Gruenewald M, et al. Non-invasive hemodynamic optimization in major abdominal surgery: a feasibility study. Minerva Anestesiol 2016; 82: 1158-69.